CLINICAL TRIAL: NCT06790680
Title: Managment of Acute Myeloid Leukemia and Myelodysplastic Patients Relapsing After Allogenic Stem Cell Transplantation: Results of the GITMO AML/MDS-relapse Registry Study
Brief Title: GITMO AML/MDS-Relapse Registry Study
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Responsible Party: Sponsor
Other Study IDs: GITMO AML/MDS-Relapse
Record Dates: First submitted 2025-01-03; First posted 2025-01-24 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukaemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The proposal arises from the increasingly pressing need to have a program of therapy for the prevention of relapse after allogeneic transplantation in patients with acute myeloid leukemia or myelodysplasia, especially if they undergo transplantation with positive minimal residual disease. These therapeutic approaches include molecular target drugs (for example, FLT-3 inhibitors when this gene lesion is present) or apoptosis inducers in combination with hypomethylating agents (for example, the combination of venetoclax and azacitidine or decitabine) or adoptive immunotherapy (for example, with infusion of donor lymphocytes).

To date, most of these therapeutic approaches are used in the phase of hematological relapse of the disease; less often they are used in the phase of persistence of minimal residual disease at the molecular level or in the phase of loss of molecular chimerism on CD34+ cells, also due to the prescribing constraints of the competent authorities (AIFA). It is believed that the collection of the Italian experience can provide important information on the use of different therapeutic platforms, in different settings. This information could be the starting point for the design of prospective and multicenter studies to be proposed in the near future.

ELIGIBILITY:
Inclusion Criteria:

* All patients with AML and MDS who underwent allo-SCT from 2015 to 2021, who relapsed and received salvage therapy for the relapse.

Exclusion Criteria:

* Patients with a diagnosis other than AML and MDS transplanted in the same period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with acute myeloid leukemia and myelodysplasia relapsed after allotransplantation and who received salvage therapy.
Sampling Method: Non-Probability Sample
Enrollment: 859 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | Through study completion, an avarage 1 year
  Complete remission rate after salvage treatment

SECONDARY OUTCOMES:
Overall survival | Through study completion, an avarage 1 year
  Secondary Outcome

CONTACTS AND LOCATIONS:
Locations (1):
- GITMO, Bologna, Italy, Italy